CLINICAL TRIAL: NCT05877963
Title: Evaluating Safety, Efficacy and Pharmacokinetics of a Modified Regimen of Ublituximab (ENHANCE )
Brief Title: Study to Evaluate Safety, Efficacy and Pharmacokinetics (PK) of a Modified Regimen of Ublituximab
Acronym: ENHANCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG1101-RMS401; 2024-519284-18-00 (Other: EU CT Number)
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ublituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Ublituximab (Experimental): Participants will receive a modified regimen of ublituximab including infusions on Day 1 of Week 1 (W1D1), Day 15, if applicable, and ublituximab 450 milligrams (mg) infusion at Week 24.
  With Protocol Version 6.0, enrollment in Part A was closed.
  Interventions: Biological: Ublituximab
- Part B: Ublituximab /Placebo (Treatment Arm A) (Experimental): Participants will receive 600 mg of ublituximab on W1D1 followed by a placebo infusion on Day 15 and 450 mg ublituximab infusion at Week 24.
  With Protocol Version 7.0, enrollment in Part B will be closed.
  Interventions: Biological: Ublituximab; Drug: Placebo
- Part B: Ublituximab (Treatment Arm B) (Experimental): Participants will receive 150 mg of ublituximab on W1D1 followed by 450 mg on Day 15 and at Week 24.
  With Protocol Version 7.0, enrollment in Part B will be closed.
  Interventions: Biological: Ublituximab
- Part C: Ublituximab (Treatment Arm C) (Experimental): Participants will receive 150 mg of ublituximab on W1D1, followed by 450 mg on Day 15 and at Week 24.
  Interventions: Biological: Ublituximab

INTERVENTIONS:
Biological: Ublituximab — Administered as an intravenous (IV) infusion.
  Other Names: TG-1101; BRIUMVI
Drug: Placebo — IV infusion
  Arms: Part B: Ublituximab /Placebo (Treatment Arm A)

SUMMARY:
The primary purpose of this phase 3b study is to assess the efficacy of a modified regimen of ublituximab in participants with relapsing multiple sclerosis (RMS) as measured by T1 Gadolinium (Gd)-enhancing lesions in Part A; PK in Part B along with efficacy of ublituximab as measured by T1 Gd-enhancing lesions in participants who had a suboptimal experience on prior anti-CD20 therapy in Part C. The study consists of 3 parts: Part A is single-armed and open-label, Part B is randomized, double-blind, placebo-controlled, and Part C is single-armed and open-label.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RMS (2017 Revised McDonald criteria).
* Participants must meet one of the following prior treatment definitions:

  1. Participants naïve to treatment.
  2. Participants previously treated with a disease modifying therapy (DMT) who have discontinued treatment prior to consent and meet the washout requirements.
* Expanded Disability Status Scale (EDSS) score ≤ 5.5 at screening.
* Neurologically stable for > 30 days prior to first dose of ublituximab.
* Female participants of childbearing potential must consent to use a medically acceptable method of contraception from consent, throughout the study period, and for 6 months after the last dose of ublituximab.
* Part C: participants currently treated with an anti-CD20 agent for at least 6 months and meet the washout requirements prior to W1D1.
* Part C: Discontinuation of current anti-CD20 must be due to suboptimal experience

Exclusion Criteria:

* History of any serious 3 Infusion Related Reaction (IRR) on prior anti-CD20 therapy.
* Primary-progressive multiple sclerosis (PPMS) or inactive Secondary Progressive MS (SPMS).
* Active chronic (or stable but treated with immune therapy) disease of the immune system other than MS (e.g., rheumatoid arthritis, scleroderma, Sjögren's syndrome, Crohn's disease, ulcerative colitis, etc.) or immunodeficiency syndrome (hereditary immune deficiency, drug-induced immune deficiency, etc.).
* Current evidence or known history of clinically significant infection, including: chronic, recurrent, or ongoing active viral, bacterial, or fungal infectious disease requiring long term systemic treatment such as, but not limited to chronic urinary tract infection, chronic pulmonary infection with bronchiectasis, tuberculosis, or active hepatitis C virus (HCV).
* Previous serious opportunistic or atypical infection.
* Evidence of chronic active or history of hepatitis B virus (HBV) infection as evidenced by a detectable hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody (HBcAb), or chronic hepatitis C infection. Participants with positive hepatitis C virus antibody (HCV Ab) are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
* History or evidence (clinical, radiological, or biomarker) of suspected or confirmed progressive multifocal leukoencephalopathy (PML).
* Receipt of any live or live-attenuated vaccines (including vaccines for varicella-zoster virus or measles) within 4 weeks prior to first study drug administration.
* Participants requiring treatment with intravenous immune globulin (IVIG) for decreased immunoglobulins within the 12 months prior to W1D1.
* Any active malignancies other than adequately treated basal, squamous cell or in situ carcinoma.
* Participants who have ever received ublituximab, alemtuzumab, cyclophosphamide, mitoxantrone, cladribine, or daclizumab (including for non-MS indications).

Note: Other Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Part A and Part C: Percentage of Participants With no Change or Reduction in Number of T1 Gd-Enhancing Lesions From Baseline to Week 48 | Baseline up to Week 48
  The Gd-enhancing T1 lesions will be evaluated using magnetic resonance imaging (MRI) technique.
Part B: Area Under the Curve Over the First 16 Weeks (AUC0-W16) of Ublituximab | Predose and at multiple timepoints up to Week 16

SECONDARY OUTCOMES:
Parts A: Percentage of Participants Free of T1 Gd-Enhancing Lesions | Week 48
  The Gd-enhancing T1 lesions will be evaluated using MRI technique.
Parts A and B: Percentage of Participants Experiencing Infusion Related Reactions (IRRs) | Up to Week 48
  IRRs are defined as infusion related adverse events (AEs) that occur within one day of an infusion and resolve within 7 days. IRRs will be reported by investigator.
Parts A: Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM-9) Scores | Part A: Baseline, Week 24 and Week 48
  The TSQM-9 is a 9-item questionnaire with 3 domains: Satisfaction, convenience, and effectiveness.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (34):
  - TG Therapeutics Investigational Trial Site, Birmingham, Alabama
  - TG Therapeutics Investigational Trial Site, Cullman, Alabama
  - TG Therapeutics Investigational Trial Site, Orange, California
  - TG Investigational Site, Fort Collins, Colorado
  - TG Therapeutics Investigational Trial Site, Washington D.C., District of Columbia
  - TG Therapeutics Investigational Trial Site, Tampa, Florida
  - TG Therapeutics Investigational Trial Site, Chicago, Illinois
  - TG Therapeutics Investigational Trial Site, Indianapolis, Indiana
  - TG Therapeutics Investigational Trial Site, Iowa City, Iowa
  - TG Therapeutics Investigational Trial Site, Overland Park, Kansas
  - TG Therapeutics Investigational Trial Site, Lutherville, Maryland
  - TG Therapeutics Investigational Trial Site, Boston, Massachusetts
  - TG Therapeutics Investigational Trial Site, Foxborough, Massachusetts
  - TG Therapeutics Investigational Trial Site, North Worcester, Massachusetts
  - TG Therapeutics Investigational Trial Site, Wellesley, Massachusetts
  - TG Investigational Site, Farmington, Michigan
  - TG Therapeutics Investigational Trial Site, Golden Valley, Minnesota
  - TG Therapeutics Investigational Trial Site, Plymouth, Minnesota
  - TG Therapeutics Investigational Trial Site, St Louis, Missouri
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial SiteCharlotte, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, Raleigh, North Carolina
  - TG Therapeutics Investigational Trial Site, Cleveland, Ohio
  - TG Therapeutics Investigational Trial Site, Dayton, Ohio
  - TG Therapeutics Investigational Trial Site, Oklahoma City, Oklahoma
  - TG Therapeutics Investigational Trial Site, Greenville, South Carolina
  - TG Therapeutics Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics Investigational Trial Site, Waco, Texas
  - TG Therapeutics Investigational Trial Site, Salt Lake City, Utah
  - TG Therapeutics Investigational Trial Site, Vienna, Virginia
  - TG Therapeutics Investigational Trial Site, Kirkland, Washington
  - TG Therapeutics Investigational Trial Site, Seattle, Washington
  - TG Therapeutics Investigational Trial Site, Spokane, Washington
  - TG Therapeutics Investigational Trial Site, Milwaukee, Wisconsin
- Poland (10):
  - TG Therapeutics Investigational Trial Site, Bydgoszcz
  - TG Therapeutics Investigational Trial Site, Katowice
  - TG Therapeutics Investigational Trial Site, Kielce
  - TG Therapeutics Investigational Trial Site, Krakow
  - TG Therapeutics Investigational Trial Site, Lodz
  - TG Therapeutics Investigational Trial Site, Olsztyn
  - TG Therapeutics Investigational Trial Site, Poznan
  - TG Therapeutics Investigational Trial Site, Warsaw
  - TG Therapeutics Investigational Trial Site, Zabrze
  - TG Therapeutics Investigational Trial Site, Żory

IPD SHARING:
Plan to Share IPD: No